CLINICAL TRIAL: NCT01699594
Title: Allergen Induced Increase in Indirect Non-allergic Bronchial Reactivity
Brief Title: Change in Airway Responsiveness After Allergen Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Saskatchewan (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: IIS-A-524; BioReb #10-227 (Other: University of Saskatchewan)
Record Dates: First submitted 2012-10-01; First posted 2012-10-03 (Estimated); Last update posted 2015-04-09 (Estimated); Status verified 2013-10

CONDITIONS: Allergic Asthma
Keywords: asthma; allergies; mannitol; methacholine
MeSH Terms: conditions — Asthma; Hypersensitivity | interventions — Mannitol; Methacholine Chloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mannitol (Experimental): This arm will assess the allergen induced change in airway responsiveness to mannitol bronchoprovocation.
  Interventions: Drug: Mannitol
- Methacholine Chloride (Active Comparator): This arm will assess the allergen induced change in airway responsiveness to methacholine bronchoprovocation.
  Interventions: Drug: Methacholine Chloride

INTERVENTIONS:
Drug: Mannitol — Indirect bronchoprovocation agent being compared to direct bronchoprovocation agent (methacholine)
  Other Names: Aridol
  Arms: Mannitol
Drug: Methacholine Chloride — Direct bronchoprovocation agent being compared to indirect bronchoprovocation agent (mannitol)
  Other Names: Provocholine
  Arms: Methacholine Chloride

SUMMARY:
Exposure to allergens changes the way the airway responds to some stimuli (methacholine). The investigators will look at whether or not exposure to allergens changes the way the airway responds to a different stimuli (mannitol) and compare that with the known stimuli (methacholine).

ELIGIBILITY:
Inclusion Criteria:

* mild, allergic asthma
* FEV1 greater than 70% predicted
* methacholine PC20 less than or equal to 16mg/ml

Exclusion Criteria:

* known sensitivity to mannitol or other excipient
* diagnosis of any other respiratory or non respiratory disease/disorder that would preclude the individual from participating
* recent thoracic, abdominal or eye surgery
* recent allergen exposure (4 weeks), respiratory infection (6 weeks)
* current immunotherapy
* pregnancy
* history of anaphylaxis
* use of asthma therapies other than short acting beta agonist

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in airway responsiveness three hours after allergen exposure | Change from Baseline at 3 hours

CONTACTS AND LOCATIONS:
Overall Officials: Donald W Cockcroft, MD, Principal Investigator — University of Saskatchewan
Locations (1):
- University of Saskatchewan, Saskatoon, Saskatchewan, Canada

REFERENCES:
- [Derived] Amakye DO, Davis BE, Martin AL, Peters GE, Cockcroft DW. Refractoriness to inhaled mannitol 3 hours after allergen challenge. Ann Allergy Asthma Immunol. 2013 Sep;111(3):182-4. doi: 10.1016/j.anai.2013.06.011. Epub 2013 Jul 12. PMID 23987192